CLINICAL TRIAL: NCT01618617
Title: Dose-response Effectiveness of 6-week Multistrain Probiotic Supplementation on Whole Gut Transit Time, Quality of Life, and Gastrointestinal Symptoms in Adults With Functional Constipation
Brief Title: Multistrain Probiotic for Functional Constipation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renew Life Formulas Inc (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 111028-SUS-REN-CTT-RA
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-06

CONDITIONS: Functional Constipation
Keywords: Constipation; Probiotic; Randomized Controlled Trial
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Probiotic, high dose (Experimental): High dose Multistrain probiotic, 100 billion cfu/day
  Interventions: Dietary Supplement: High dose Multistrain probiotic, 100 billion cfu/day
- Probiotic, low dose (Experimental): Low dose Multistrain probiotic, 15 billion cfu/day
  Interventions: Dietary Supplement: Low dose Multistrain probiotic, 15 billion cfu/day
- Placebo (Placebo Comparator): Placebo

INTERVENTIONS:
Dietary Supplement: High dose Multistrain probiotic, 100 billion cfu/day — 100 billion cfu live bacteria (60 billion cfu bifidobacterium cultures and 40 billion lactobacillus cultures).
  Other Names: Ultimate Flora Critical
  Arms: Probiotic, high dose
Dietary Supplement: Low dose Multistrain probiotic, 15 billion cfu/day — 15 billion cfu live bacteria (9 billion cfu bifidobacterium cultures and 6 billion lactobacillus cultures).
  Other Names: Ultimate Flora Critical Care capsules
  Arms: Probiotic, low dose

SUMMARY:
Subjects will be screened and will enter a placebo-only 2-week run-in period during which constipation symptoms will be evaluated and any disallowed products (e.g. probiotics) must be discontinued. Following successful completion of the run-in period, subjects will be randomized to probiotic (high or low-dose groups) or placebo. Subjects will then consume their assigned product daily for 6 weeks. Subjects will undergo abdominal x-rays on study days 0 and 42 to assess transit time with each examination preceded by 6 days of radiopaque Sitz marker ingestion. Subject diaries will be used to collect bowel movement frequency, stool consistency, concomitant medications, and adverse events each day during the trial. Stool samples will be collected at baseline and end of study to assess fecal probiotic count. PAC-QOL, WCS, and GSRS questionnaires will be administered at baseline and day 42. 24-hour food recalls will be administered at day 0 and 42 and the following parameters will be assessed: total calories, carbohydrate, fat, protein, fiber, and liquid intake. Weekly physical activity recalls will be completed.

DETAILED DESCRIPTION:
Primary Endpoint: Whole gut transit time

The primary endpoint of this clinical trial is whole gut transit time, which will be assessed using abdominal x-rays (supine anteroposterior kidney-ureter-bladder, KUB) on days 0 and 42. Each subject will ingest 24 radiopaque Sitz markers each day for 6 consecutive days at the same time of the day prior to abdominal x-rays on days 0 and 42, also taken at the same time of the day that the markers were taken. The number of markers present in the right, left, and rectosigmoid colon will be summed to yield a total marker count. Whole gut transit time will be calculated using the classic film estimate as described in the following formula:

WGTT = ni x (t/N) 19, 20

where ni is the number of markers observed on x-ray, t is the time between marker ingestions in hours, and N is the total number of markers ingested each day. Thus, in this study, t/N equals 1 (24 markers per capsule/24 hours between marker ingestions), and WGTT is, therefore, equal to the total marker count 19, 20.

Marker counts will be identified by a single radiologist at each site who will remain blinded to subject treatment assignment.

The methodology above is safe, noninvasive, and the two abdominal x-rays required for this study collectively expose each subject to radiation doses of approximately 140 millirem (equivalent to 1.4 millisievert). The overall lifetime risk that this radiation dosage may cause cancer is approximately 1 in 4,000 for women aged 18 years, 1 in 6,000 for men aged 18 years, 1 in 20,000 for women aged 70 years, and 1 in 25,000 for men aged 70 years. Similar abdominal x-ray methodology has been utilized in similar studies in adults aged 18 years and older 21, 22.

Secondary Endpoint: Patient Assessment of Constipation Quality of Life (PAC-QoL) The PAC-QoL (Appendix A) is a 28-question survey that measures the impact that constipation has on daily life over the past 2 weeks. The questions are comprised of four subscales (worries and concerns, physical discomfort, psychosocial discomfort, and satisfaction) and an overall scale. Multinational studies have demonstrated that the PAC-QoL is internally consistent, reproducible, valid, and responsive to improvements over time 23. Subjects will complete the PAC-QoL at days 0 and 42.

Secondary Endpoint: Wexner Constipation Score (WCS) The Wexner Constipation Score (WCS) (Appendix B) is an 8-question survey that assesses frequency of bowel movements, straining, incomplete evacuation, abdominal pain, time needed for defecation, assistance for defecation, unsuccessful attempts, and duration of constipation. The WCS is a validated questionnaire since WCS scores correlate well with objective physiologic findings in constipated patients 24. Subjects will complete the WCS at days 0 and 42.

Secondary Endpoint: Gastrointestinal Symptom Rating Scale (GSRS) The GSRS (Appendix C) is a 15-item instrument designed to assess common GI symptoms 25. It has five subscales (reflux, diarrhea, constipation, indigestion, and abdominal pain) with subscale scores ranging from 1 (no discomfort) to 7 (severe discomfort). Higher scores represent higher symptom burden. Subjects will complete the GSRS at days 0 and 42.

Secondary Endpoint: Stool frequency Throughout the study, subjects will record the number of defecations per day in a diary throughout the study. The stool frequency endpoint will be the absolute change in weekly stools in each group from the second week of the run-in period to the sixth study week.

Secondary Endpoint: Stool Consistency Stool consistency will be rated with the Bristol Stool Scale Form 26 (Appendix D). Subjects will grade each stool using a daily diary throughout the study. The stool consistency endpoint will be the mean change in each group from the second week of the run-in period to the sixth study week.

Secondary Endpoint: Fecal Probiotic Count Stool samples will be collected at baseline and end of study to assess fecal probiotic count via live culture, which will include total lactobacillis count and total bifidobacterium count. At the Day 0 visit following randomization, subjects will be provided two separate stool collection kits-one to be used at baseline and one to be used at the end of the supplementation period.

After receipt of the kits, subjects must provide the first stool sample before taking the first dose of study product, regardless of the length of time needed to have a bowel movement. The stool sample can be provided at the study site on Day 0 or the subject may collect their first stool thereafter and ship the sample in a provided refrigerated container to the laboratory for analysis. Once the first stool sample is provided, the subject may then begin consuming study product.

During the final 3 days of the supplementation period (i.e. Day 40, 41, or 42), subjects must provide another stool sample and ship the sample in a provided refrigerated container to the laboratory for analysis. This must be completed before returning to the site for the Day 42 assessments.

Secondary Endpoint: Adverse Events Adverse events (AEs) will be assessed throughout this clinical study. The main safety endpoint will be the proportion of subjects in each group that report one of more AEs at any time during the study. Please see Section 6 for additional details on the AE assessment.

Ancillary Outcome: International Physical Activity Questionnaire (IPAQ)-short version The International Physical Activity Questionnaire (IPAQ)-short version is a validated questionnaire suitable for quantifying physical activity levels in adults (Appendix E) 27.

Ancillary Outcome: 24-hour Food Recall A 24-hour food recall will be completed in order to quantify total calories, carbohydrate (g), fat (g), protein (g), fiber (g), and liquid intake (ml). The food recall must take place on a weekday (Monday through Thursday). Subjects must record all foods and beverages consumed as well as the quantity of each (recorded as weight or volume).

Ancillary Outcome: Concomitant medication use Throughout the study, subjects will record use of any concomitant medication and, if required, the need for rescue medication each day in a diary.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years
2. Body mass index 18.5 to 39.9 kg/m2
3. Meets the criteria below over the last 3 months with symptom onset at least 6 months prior (Rome III definition of functional constipation 1):

   * Meets 2 or more of the following criteria:

     * Straining during at least 25% of defecations
     * Lumpy or hard stools in at least 25% of defecations
     * Sensation of incomplete evacuation for at least 25% of defecations
     * Sensation of anorectal obstruction/blockage for at least 25% of defecations
     * Manual maneuvers to facilitate at least 25% of defecations (e.g. digital evacuation, support of the pelvic floor)
     * Fewer than three defecations per week
   * Loose stools are rarely present without the use of laxatives
   * Insufficient criteria for irritable bowel syndrome
4. Agree to use contraception throughout study period, unless postmenopausal or surgically sterile (females only)
5. Able to understand the nature and purpose of the study including potential risks and side effects
6. Willing to consent to study participation and to comply with study requirements
7. Successful completion of 2-week run-in period, defined as:

   * Must meet the Rome III definition of functional constipation during this 2-week period
   * Completion of all study-related questionnaires

Exclusion Criteria:

1. Major gastrointestinal complication (e.g. Crohn's disease, ulcer, cancer)
2. Prior abdominal surgery that, in the investigator's opinion, may confound study outcomes
3. Clinically significant systemic disease (e.g. cancer, diabetes, CAD)
4. Consumption of probiotics or prebiotics within 2 weeks of randomization
5. Antibiotic use within 4 weeks of randomization
6. Laxative or other constipation medication use within 2 weeks of randomization
7. Eating disorder
8. Known allergies to any substance in the study product, including lactose intolerance
9. Pregnant or breastfeeding women
10. History of alcohol, drug, or medication abuse
11. Participation in another study with any investigational product within 3 months of randomization
12. Any condition that could, in the opinion of the investigator, preclude the subject's ability to successfully and safely complete the study or that may confound study outcomes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Whole gut transit time | 6 weeks

SECONDARY OUTCOMES:
Patient Assessment of Constipation Quality of Life (PAC-QOL) | 6 weeks
Wexner Constipation Score (WCS) | 6 weeks
Gastrointestinal Symptom Rating Scale (GSRS) | 6 weeks
Stool frequency | 6 weeks
Stool consistency | 6 weeks
Fecal probiotic count | 6 weeks
Adverse events | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn Hattner, MPH, RD, Principal Investigator — Stanford University
Locations (1):
- Sprim, San Francisco, California, United States